CLINICAL TRIAL: NCT00435708
Title: Effect of Increased Fruit and Vegetable Intake on Airway Inflammation and Oxidative Stress in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effect of Increased Fruit and Vegetable Intake on Chronic Obstructive Pulmonary Disease (COPD)
Acronym: DISCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Michelle McKinley, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ref 200651
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Fruit; Vegetables; Oxidative stress; Inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low fruit and vegetables (No Intervention): Control - two or less portions fruit and vegetables/day
- High fruit and vegetables (Experimental): 5 portions fruit and vegetables/day
  Interventions: Behavioral: 5 portions fruit and vegetables/day

INTERVENTIONS:
Behavioral: 5 portions fruit and vegetables/day — Participants consume > = 5 portions fruit and veg per day
  Arms: High fruit and vegetables

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the UK's fastest growing fatal disease and is estimated to cost the health service close to £1 billion every year. Around 80,000 people in Northern Ireland suffer from COPD. COPD is clinically defined as a slowly progressive condition characterised by airflow limitation, which is largely irreversible. Chronic inflammation and oxidative stress are key components of the underlying pathological process resulting in airflow limitation. Dietary factors and nutrients that have antioxidant or anti-inflammatory properties are therefore of interest with respect to the aetiology of COPD. The antioxidant vitamins C, E and beta-carotene are all present in the lung milieu. Such antioxidants represent the lung's first line of defence against oxygen free radicals. Observational studies indicate that a low dietary intake of antioxidant nutrients, or foods rich in antioxidants (e.g. fruit and vegetables), is associated with decreased lung function and increased risk of COPD. To date, there have been no food-based dietary interventions investigating the effect of increased fruit and vegetable intake on COPD. The investigators propose to recruit people with mild to moderate COPD and low fruit and vegetable intakes (<=2 portions daily) and randomise them to one of two study arms for 12 weeks - either to increase fruit and vegetable consumption to at least 5 portions a day, or to follow their normal diet. Airway and systemic oxidative stress and inflammation will be assessed at baseline and post-intervention in order to determine if fruit and vegetables have the potential to alleviate the oxidative stress and airway inflammation associated with COPD.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe COPD (according to GOLD classification)
* oxygen saturation >= 92 KPa
* symptomatically stable
* habitually low fruit and vegetable intakes (<=2 portions daily)
* exercise limited by shortness of breath (rather than e.g. angina, arthritis)

Exclusion Criteria:

* diabetes
* taking antioxidant supplements or drugs
* oxygen saturation <8KPa

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Young, MD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University Belfast, Belfast, Co.Antrim, United Kingdom

REFERENCES:
- [Result] Baldrick FR, Elborn JS, Woodside JV, Treacy K, Bradley JM, Patterson CC, Schock BC, Ennis M, Young IS, McKinley MC. Effect of fruit and vegetable intake on oxidative stress and inflammation in COPD: a randomised controlled trial. Eur Respir J. 2012 Jun;39(6):1377-84. doi: 10.1183/09031936.00086011. Epub 2011 Nov 16. PMID 22088966

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Control: Control -two or fewer portions fruit and vegetables/day
- 2 Intervention: 5 portions fruit and vegetables/day
  5 portions fruit and vegetables/day: Participants consume > = 5 portions fruit and veg per day
Period: Overall Study
Arm/Group | 1 Control | 2 Intervention
Started | 41 | 40
Completed | 37 | 38
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Low FV Group: Control - two or less portions fruit and vegetables/day
- High FV Group: 5 portions fruit and vegetables/day
  5 portions fruit and vegetables/day: Participants consume > = 5 portions fruit and veg per day
- Total: Total of all reporting groups
Arm/Group | Low FV Group | High FV Group | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.3) | 63.2 (9.1) | 62.2 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 25 | 21 | 46
Region of Enrollment [Number; unit: participants]
  United Kingdom | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Intake of Fruit and Vegetables (Number of Portions Per Day);
Description: A series of 7-day diet histories were completed by each participant at weeks 0 and 12 in order to assess baseline diet and self-reported compliance with the intervention; average daily FV intake was then hand-counted from these records;
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Portions per day
Groups:
- Control: Control -two or fewer portions fruit and vegetables/day
- Intervention: 5 portions fruit and vegetables/day
  5 portions fruit and vegetables/day: Participants consume > = 5 portions fruit and veg per day
Arm/Group | Control | Intervention
Number analyzed (Participants) | 41 | 40
Portions per day | 1.9 (0.5) | 6.1 (1.8)

2. Primary Outcome: Markers of Airway Inflammation in Induced Sputum - Sputum 8-isoprostane
Description: Markers of Airway Inflammation in Induced Sputum - Sputum 8-isoprostane ng/ml
Time Frame: 12 Weeks
Measure: Geometric Mean (Inter-Quartile Range); unit: ng/ml
Arm/Group | Low Fruit and Vegetables | High Fruit and Vegetables
Number analyzed (Participants) | 27 | 25
ng/ml | 1.70 [1.26 to 2.42] | 1.83 [1.18 to 2.63]

3. Secondary Outcome: Biochemical Markers of Nutritional Status Plasma Vitamin C
Description: Plasma vitamin C concentration umol/L
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: umol/l
Arm/Group | Low FV Group | High FV Group
Number analyzed (Participants) | 36 | 38
umol/l | 33.44 (21.19) | 47.64 (19.23)

ADVERSE EVENTS:
Time Frame: Baseline, 6 week, 12 week
Arm/Group | 1 Control | 2 Intervention
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 0/41 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes